CLINICAL TRIAL: NCT02252172
Title: A Phase 3 Study Comparing Daratumumab, Lenalidomide, and Dexamethasone (DRd) vs Lenalidomide and Dexamethasone (Rd) in Subjects With Previously Untreated Multiple Myeloma Who Are Ineligible for High Dose Therapy
Brief Title: Study Comparing Daratumumab, Lenalidomide, and Dexamethasone With Lenalidomide and Dexamethasone in Participants With Previously Untreated Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR104762; 54767414MMY3008 (Other: Janssen Research & Development, LLC); 2014-002273-11 (EudraCT Number)
Record Dates: First submitted 2014-08-11; First posted 2014-09-30 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Daratumumab; JNJ-54767414; Lenalidomide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lenalidomide and Dexamethasone (Rd) (Active Comparator): Participants will receive Lenalidomide 25 mg capsule orally on Day 1 through Day 21 of each 28-day cycle, Dexamethasone 40 mg orally or intravenously once a week. Study treatment continues until disease progression, unacceptable toxicity, or end of study (maximum up to 7 years after last subject is randomized) whichever comes first.
  Interventions: Drug: Daratumumab IV; Drug: Lenalidomide; Drug: Dexamethasone
- Daratumumab + Lenalidomide + Dexamethasone (DRd) (Active Comparator): Participants will receive Daratumumab 16 milligram per kilogram (mg/kg) by intravenous infusion, once a week for 8 weeks, then once every other week for 16 weeks, thereafter once every 4 weeks, Lenalidomide 25 mg capsule orally on Day 1 through Day 21 of each 28-day cycle, Dexamethasone 40 mg orally or intravenously once a week. Following implementation of protocol amendment 8, participants still receiving treatment with daratumumab IV will have the option to switch to daratumumab SC on Day 1 of any cycle, at the discretion of the investigator. Daratumumab subcutaneous (SC) will be administered by SC injection at a fixed dose of 1800 mg once every 4 weeks until documented progression, unacceptable toxicity, or study completion. Study treatment continues until disease progression, unacceptable toxicity, or end of study (maximum up to 7 years after last subject is randomized) whichever comes first.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Drug: Daratumumab SC

INTERVENTIONS:
Drug: Daratumumab IV — Daratumumab will be administered at a dose of 16 milligram per kilogram (mg/kg) by intravenous (IV) infusion, once a week for 8 weeks, then once every other week for 16 weeks, thereafter once every 4 weeks until documented progression of disease, unacceptable toxicity, or end of study (maximum up to 7 years).
  Other Names: JNJ-54767414
  Arms: Lenalidomide and Dexamethasone (Rd)
Drug: Lenalidomide — Lenalidomide 25 mg capsule orally on Day 1 through Day 21 of each 28-day cycle.
Drug: Dexamethasone — Dexamethasone 40 mg orally or intravenously once in a week.
Drug: Daratumumab SC — Daratumumab SC will be administered by SC injection at a fixed dose of 1800 mg once every 4 weeks until documented progression, unacceptable toxicity, or study end. Following implementation of protocol amendment 8, participants still receiving treatment with daratumumab IV will have the option to switch to daratumumab SC on Day 1 of any cycle, at the discretion of the investigator.
  Other Names: JNJ-54767414
  Arms: Daratumumab + Lenalidomide + Dexamethasone (DRd)

SUMMARY:
The purpose of this study is to compare the efficacy of daratumumab in combination with lenalidomide and dexamethasone to that of lenalidomide and dexamethasone in terms of progression-free survival (PFS) in participants with newly diagnosed multiple myeloma (a blood cancer of plasma cells) who are not candidates for high dose chemotherapy (treatment of disease, usually cancer, by chemical agents) and autologous stem cell transplant (ASCT).

DETAILED DESCRIPTION:
This is a Phase 3, randomized (study drug assigned by chance), open-label (participants and researchers are aware about the treatment, participants are receiving), active-controlled (study in which the experimental treatment or procedure is compared to a standard treatment or procedure), parallel-group (each group of participants will be treated at the same time), and multicenter (when more than one hospital or medical school team work on a medical research study) study in participants with newly diagnosed multiple myeloma and who are not candidates for high dose chemotherapy and ASCT. All the eligible participants will be randomly assigned to receive either lenalidomide and dexamethasone (Rd) (Arm A) or daratumumab in combination with lenalidomide and dexamethasone (DRd) (Arm B). Daratumumab (16 milligram per kilogram [mg/kg]) will be administered weekly for first 8 weeks (Cycles 1 to 2) of treatment and then every other week for 16 weeks (Cycles 3 to 6), then every 4 weeks (from Cycle 7 and beyond) until progression of disease or unacceptable toxicity. Lenalidomide will be administered at a dose of 25 mg orally on Days 1 through 21 of each 28-day cycle, and dexamethasone will be administered at a dose of 40 mg once a week for both treatment arms. Participants in both treatment arms will continue lenalidomide and dexamethasone until disease progression or unacceptable toxicity. All participants randomized to Treatment Arm B (DRd) in this study initially received daratumumab IV formulation; however, following implementation of protocol amendment 8, participants still receiving treatment with daratumumab IV will have the option to switch to daratumumab SC on Day 1 of any cycle, at the discretion of the investigator. Daratumumab subcutaneous (SC) will be administered by SC injection at a fixed dose of 1800 mg once every 4 weeks until documented progression, unacceptable toxicity, or study completion. Participants in Arm A who have sponsor-confirmed disease progression may have the option to receive daratumumab provided by the sponsor (in any subsequent line of therapy) in the Follow-up phase. The study consists of 3 phases: Screening Phase (within 21 days prior to the first dose administration on Day 1), Treatment Phase (Day 1 up to discontinuation of all study treatment), and Follow-up Phase (from discontinuation of all study treatment up to death, lost to follow up, consent withdrawal, or study end, whichever occurs first). The maximum duration of study will be 7 years after last participant is randomized. Efficacy will primarily be evaluated by PFS. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have documented multiple myeloma satisfying the CRAB (calcium elevation, renal insufficiency, anemia and bone abnormalities) criteria, monoclonal plasma cells in the bone marrow greater than or equal to (>=) 10 percent (%) or presence of a biopsy proven plasmacytoma and measurable disease as defined by any of the following: (a) immunoglobulin (Ig) G myeloma (serum monoclonal paraprotein [M-protein] level >=1.0 gram/deciliter [g/dL] or urine M-protein level >=200 milligram[mg]/24 hours[hrs]; or (b) IgA, IgM, IgD, or IgE multiple myeloma (serum M-protein level >=0.5 g/dL or urine M-protein level >=200 mg/24 hrs); or (c) light chain multiple myeloma without measurable disease in serum or urine (serum immunoglobulin free light chain >=10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio)
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Participants who are newly diagnosed and not considered for high-dose chemotherapy due to: being age >=65 years; or participants less than (<) 65 years with presence of important comorbid condition(s) likely to have a negative impact on tolerability of high dose chemotherapy with stem cell transplantation. Sponsor review and approval of participants below 65 years of age is required before randomization
* Women of childbearing potential must commit to either abstain continuously from sexual intercourse or to use 2 methods of reliable birth control simultaneously as deemed appropriate by the Investigator. Contraception must begin 4 weeks prior to dosing and must continue for 3 months after the last dose of daratumumab
* Man, who is sexually active with a woman of child-bearing potential must agree to use a latex or synthetic condom, even if he had a successful vasectomy, must agree to use an adequate contraception method as deemed appropriate by the Investigator, and must also agree to not donate sperm during the study and for 4 weeks after last dose of lenalidomide and 4 months after last dose of daratumumab

Exclusion Criteria:

* Participant has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance (presence of serum M-protein <3 g/dL; absence of lytic bone lesions, anemia, hypercalcemia, and renal insufficiency related to the M-protein), or smoldering multiple myeloma (asymptomatic multiple myeloma with absence of related organ or tissue impairment end organ damage)
* Participant has a diagnosis of Waldenström's disease, or other conditions in which IgM M protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions
* Participant has a history of malignancy (other than multiple myeloma) within 5 years before the date of randomization (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the Investigator, with concurrence with the Sponsor's medical monitor, is considered cured with minimal risk of recurrence within 5 years)
* Participant has prior or current systemic therapy or SCT for multiple myeloma, with the exception of an emergency use of a short course (equivalent of dexamethasone 40 mg/day for 4 days) of corticosteroids before treatment
* Participant has had radiation therapy within 14 days of randomization
* Participant has known chronic obstructive pulmonary disease (COPD) (defined as a forced expiratory volume in 1 second [FEV1] <50% of predicted normal), persistent asthma, or a history of asthma within the last 2 years (controlled intermittent asthma or controlled mild persistent asthma is allowed)
* Participants with known or suspected COPD must have a FEV1 test during Screening
* Participant is known to be seropositive for human immunodeficiency virus (HIV) or hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg] or antibodies to hepatitis B surface and core antigens [anti-HBs and anti-HBc, respectively]) or hepatitis C (anti-HCV antibody positive or HCV-ribonucleic acid [RNA] quantitation positive)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 737 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2024-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (206):
- United States (83):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Glendale, Arizona
  - Berkeley, California
  - Beverly Hills, California
  - El Cajon, California
  - Greenbrae, California
  - Los Angeles, California
  - Oceanside, California
  - San Diego, California
  - West Hills, California
  - Whittier, California
  - Denver, Colorado
  - Fort Collins, Colorado
  - Glenwood Springs, Colorado
  - New Haven, Connecticut
  - Norwalk, Connecticut
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Boynton Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Lake City, Florida
  - St. Petersburg, Florida
  - Weston, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Macon, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Niles, Illinois
  - Fort Wayne, Indiana
  - Iowa City, Iowa
  - Louisville, Kentucky
  - Lafayette, Louisiana
  - Marrero, Louisiana
  - Shreveport, Louisiana
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Frederick, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Duluth, Minnesota
  - Rochester, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Hooksett, New Hampshire
  - Brick, New Jersey
  - Hackensack, New Jersey
  - Livingston, New Jersey
  - Plainfield, New Jersey
  - Summit, New Jersey
  - Mineola, New York
  - New York, New York
  - Rochester, New York
  - Asheboro, North Carolina
  - Charlotte, North Carolina
  - Pinehurst, North Carolina
  - Winston-Salem, North Carolina
  - Canton, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Bend, Oregon
  - Bethlehem, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Spartanburg, South Carolina
  - Sioux Falls, South Dakota
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Edinburg, Texas
  - Fort Sam Houston, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Ogden, Utah
  - Seattle, Washington
  - Spokane, Washington
  - Tacoma, Washington
- Australia (9):
  - Box Hill
  - Fitzroy
  - Footscray
  - Kogarah
  - Kurralta Park
  - Nedlands
  - New South Wales
  - Woodville
  - Woolloongabba
- Austria (5):
  - Innsbruck
  - Linz
  - Salzburg
  - Vienna
  - Wien Wien
- Belgium (5):
  - Bruges
  - Brussels
  - Haine Saint Paul La Louviere
  - Leuven
  - Liège
- Canada (7):
  - Calgary, Alberta
  - Nova Scotia, Nova Scotia
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - N/a N/a
- Denmark (3):
  - Aarhus C
  - Odense
  - Vejle
- France (41):
  - Amiens N/a Picardie
  - Angers
  - Bayonne
  - Bretagne
  - Caen
  - Cergy-Pontoise
  - Chalon-sur-Saône
  - Clermont-Ferrand
  - Créteil
  - Dijon
  - Dunkirk
  - Grenoble
  - La Roche-sur-Yon
  - Le Chesnay
  - Le Mans
  - Lille
  - Limoges
  - Lyon
  - Marseille
  - Metz-Tessy
  - Montivilliers
  - Montpellier
  - Mulhouse
  - Nantes
  - Nice
  - Paris
  - Perpignan
  - Pessac
  - Périgueux
  - Poitiers
  - Reims
  - Rennes
  - Rouen
  - Saint-Brieuc
  - Saint-Priest-en-Jarez
  - Saint-Quentin
  - St-Malo
  - Strasbourg
  - Toulouse
  - Tours
  - Vandœuvre-lès-Nancy
- Germany (20):
  - Aschaffenburg
  - Bad Berka
  - Bonn
  - Braunschweig
  - Dresden
  - Essen
  - Frankfurt
  - Hanover
  - Heidelberg
  - Hessen
  - Kiel
  - Koblenz
  - Mainz
  - Mannheim
  - Rostock
  - Schwerin
  - Stuttgart
  - Tübingen
  - Ulm
  - Villingen-Schwenningen
- Ireland (2):
  - Dublin
  - Galway
- Israel (6):
  - Hadera
  - Haifa
  - Jerusalem
  - Nahariya
  - Petah Tikva
  - Tel Aviv
- Netherlands (4):
  - Hilversum
  - Hoofddorp
  - Rotterdam
  - Tilburg
- Sweden (9):
  - Falun
  - Gothenburg
  - Halmstad
  - Helsingborg
  - Huddinge
  - Luleå
  - Lund
  - Örebro
  - Stockholm
- United Kingdom (12):
  - Aberdeen
  - Canterbury
  - Dundee
  - Leeds
  - London
  - Manchester
  - Nottingham
  - Oxford
  - Plymouth
  - Southampton
  - Truro
  - Wolverhampton

REFERENCES:
- [Derived] Perrot A, Facon T, Plesner T, Usmani SZ, Kumar S, Bahlis NJ, Hulin C, Orlowski RZ, Nahi H, Mollee P, Ramasamy K, Roussel M, Jaccard A, Delforge M, Karlin L, Arnulf B, Chari A, Wang G, Gupta-Werner N, Kaila S, Pei H, Matt K, Gries KS, Carson R, Borgsten F, Weisel K. Sustained Improvement in Health-Related Quality of Life in Transplant-Ineligible Newly Diagnosed Multiple Myeloma Treated With Daratumumab, Lenalidomide, and Dexamethasone: MAIA Final Analysis of Patient-Reported Outcomes. Eur J Haematol. 2025 May;114(5):883-889. doi: 10.1111/ejh.14392. Epub 2025 Feb 14. PMID 39952901
- [Derived] Moreau P, Facon T, Usmani SZ, Bahlis N, Raje N, Plesner T, Orlowski RZ, Basu S, Nahi H, Hulin C, Quach H, Goldschmidt H, O'Dwyer M, Perrot A, Venner CP, Weisel K, Tiab M, Macro M, Frenzel L, Leleu X, Wang G, Pei H, Krevvata M, Carson R, Borgsten F, Kumar SK. Daratumumab plus lenalidomide/dexamethasone in untreated multiple myeloma: analysis of key subgroups of the MAIA study. Leukemia. 2025 Mar;39(3):710-719. doi: 10.1038/s41375-024-02506-1. Epub 2025 Jan 15. PMID 39815052
- [Derived] Almansour SA, Alqudah MAY, Abuhelwa Z, Al-Shamsi HO, Alhuraiji A, Semreen MH, Bustanji Y, Alzoubi KH, Modi ND, Mckinnon RA, Sorich MJ, Hopkins AM, Abuhelwa AY. Antithrombotic utilization, adverse events, and associations with treatment outcomes in multiple myeloma: pooled analysis of three clinical trials. Ther Adv Med Oncol. 2024 Sep 2;16:17588359241275387. doi: 10.1177/17588359241275387. eCollection 2024. PMID 39229471
- [Derived] Facon T, Kumar SK, Plesner T, Orlowski RZ, Moreau P, Bahlis N, Basu S, Nahi H, Hulin C, Quach H, Goldschmidt H, Perrot A, Weisel K, Raje N, Macro M, Frenzel L, Leleu X, Wang J, Rampelbergh RV, Uhlar CM, Vermeulen J, Duran J, Borgsten F, Usmani SZ. Plain language summary of the MAIA study of daratumumab plus lenalidomide and dexamethasone for the treatment of people with newly diagnosed multiple myeloma. Future Oncol. 2023 Apr;19(13):887-895. doi: 10.2217/fon-2023-0082. Epub 2023 May 22. PMID 37212642
- [Derived] Mateos MV, Rigaudeau S, Basu S, Spicka I, Schots R, Wrobel T, Cook G, Beksac M, Gries KS, Kudva A, Tromp B, Van Rampelbergh R, Pei H, Wroblewski S, Carson R, Delioukina M, White D. Switching to daratumumab SC from IV is safe and preferred by patients with multiple myeloma. J Oncol Pharm Pract. 2023 Jul;29(5):1172-1177. doi: 10.1177/10781552221103551. Epub 2022 Sep 6. PMID 36067063
- [Derived] Facon T, Kumar SK, Plesner T, Orlowski RZ, Moreau P, Bahlis N, Basu S, Nahi H, Hulin C, Quach H, Goldschmidt H, O'Dwyer M, Perrot A, Venner CP, Weisel K, Mace JR, Raje N, Tiab M, Macro M, Frenzel L, Leleu X, Ahmadi T, Wang J, Van Rampelbergh R, Uhlar CM, Tromp B, Delioukina M, Vermeulen J, Usmani SZ. Daratumumab, lenalidomide, and dexamethasone versus lenalidomide and dexamethasone alone in newly diagnosed multiple myeloma (MAIA): overall survival results from a randomised, open-label, phase 3 trial. Lancet Oncol. 2021 Nov;22(11):1582-1596. doi: 10.1016/S1470-2045(21)00466-6. Epub 2021 Oct 13. PMID 34655533
- [Derived] Cavo M, San-Miguel J, Usmani SZ, Weisel K, Dimopoulos MA, Avet-Loiseau H, Paiva B, Bahlis NJ, Plesner T, Hungria V, Moreau P, Mateos MV, Perrot A, Iida S, Facon T, Kumar S, van de Donk NWCJ, Sonneveld P, Spencer A, Krevvata M, Heuck C, Wang J, Ukropec J, Kobos R, Sun S, Qi M, Munshi N. Prognostic value of minimal residual disease negativity in myeloma: combined analysis of POLLUX, CASTOR, ALCYONE, and MAIA. Blood. 2022 Feb 10;139(6):835-844. doi: 10.1182/blood.2021011101. PMID 34289038
- [Derived] San-Miguel J, Avet-Loiseau H, Paiva B, Kumar S, Dimopoulos MA, Facon T, Mateos MV, Touzeau C, Jakubowiak A, Usmani SZ, Cook G, Cavo M, Quach H, Ukropec J, Ramaswami P, Pei H, Qi M, Sun S, Wang J, Krevvata M, DeAngelis N, Heuck C, Van Rampelbergh R, Kudva A, Kobos R, Qi M, Bahlis NJ. Sustained minimal residual disease negativity in newly diagnosed multiple myeloma and the impact of daratumumab in MAIA and ALCYONE. Blood. 2022 Jan 27;139(4):492-501. doi: 10.1182/blood.2020010439. PMID 34269818
- [Derived] Perrot A, Facon T, Plesner T, Usmani SZ, Kumar S, Bahlis NJ, Hulin C, Orlowski RZ, Nahi H, Mollee P, Ramasamy K, Roussel M, Jaccard A, Delforge M, Karlin L, Arnulf B, Chari A, He J, Ho KF, Van Rampelbergh R, Uhlar CM, Wang J, Kobos R, Gries KS, Fastenau J, Weisel K. Health-Related Quality of Life in Transplant-Ineligible Patients With Newly Diagnosed Multiple Myeloma: Findings From the Phase III MAIA Trial. J Clin Oncol. 2021 Jan 20;39(3):227-237. doi: 10.1200/JCO.20.01370. Epub 2020 Dec 16. PMID 33326255
- [Derived] Facon T, Kumar S, Plesner T, Orlowski RZ, Moreau P, Bahlis N, Basu S, Nahi H, Hulin C, Quach H, Goldschmidt H, O'Dwyer M, Perrot A, Venner CP, Weisel K, Mace JR, Raje N, Attal M, Tiab M, Macro M, Frenzel L, Leleu X, Ahmadi T, Chiu C, Wang J, Van Rampelbergh R, Uhlar CM, Kobos R, Qi M, Usmani SZ; MAIA Trial Investigators. Daratumumab plus Lenalidomide and Dexamethasone for Untreated Myeloma. N Engl J Med. 2019 May 30;380(22):2104-2115. doi: 10.1056/NEJMoa1817249. PMID 31141632

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenalidomide + Dexamethasone (Rd): Participants received Lenalidomide 25 milligrams (mg) capsule orally daily on Day 1 through Day 21 of each 28-day cycle, Dexamethasone 40 mg orally or intravenously (IV) once a week (QW) until disease progression or unacceptable toxicity up to 77.5 months. After completion of treatment, participants entered follow-up phase and were not started on subsequent anti-myeloma therapy without confirmed disease progression (assessed by the International Myeloma Working Group [IMWG] criteria).
- Daratumumab + Lenalidomide + Dexamethasone (DRd): Participants received Daratumumab 16 milligrams per kilograms (mg/kg) IV QW for the first 8 weeks (cycles 1-2) and then every 2 weeks (Q2W) for 16 weeks (Cycle 3-6), then every 4 weeks (Q4W) (from Cycle 7 and beyond) (each cycle of 28 days), Lenalidomide 25 mg capsule orally daily on Day 1 through Day 21 of each 28-day cycle, Dexamethasone 40 mg orally or IV QW until disease progression or unacceptable toxicity up to 77.3 months. After implementation of Amendment 8, participants who were ongoing with daratumumab IV treatment were given an option to switch to daratumumab subcutaneous (SC) injection on Day 1 of any cycle, as per investigator's discretion. After completion of treatment, participants entered follow-up phase and were not started on subsequent anti-myeloma therapy without confirmed disease progression (assessed by IMWG criteria).
Period: Overall Study
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Started | 369 | 368
Treated | 365 | 364
Completed | 0 | 0
Not Completed | 369 | 368
Not completed — Lost to Follow-up | 9 | 6
Not completed — Death | 218 | 175
Not completed — Withdrawal by Subject | 20 | 15
Not completed — Physician Decision | 0 | 1
Not completed — End of data collection | 122 | 170
Not completed — Site closure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd) | Total
Number analyzed (Participants) | 369 | 368 | 737
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.2 (5.66) | 74.0 (5.44) | 74.1 (5.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 179 | 353
  Male | 195 | 189 | 384
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 23
  Not Hispanic or Latino | 352 | 347 | 699
  Unknown or Not Reported | 5 | 10 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 339 | 336 | 675
  Black or African American | 16 | 12 | 28
  Asian | 2 | 3 | 5
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  Other | 6 | 6 | 12
  Unknown | 1 | 2 | 3
  Not Reported | 4 | 9 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 18 | 17 | 35
  Austria | 11 | 3 | 14
  Belgium | 5 | 2 | 7
  Canada | 28 | 24 | 52
  Denmark | 6 | 10 | 16
  France | 155 | 157 | 312
  Germany | 16 | 19 | 35
  Ireland | 3 | 4 | 7
  Israel | 3 | 5 | 8
  Italy | 3 | 3 | 6
  Netherlands | 1 | 4 | 5
  Sweden | 12 | 10 | 22
  United Kingdom | 34 | 33 | 67
  United States | 74 | 77 | 151
Stage of Disease (ISS) [Count of Participants; unit: Participants] — The International Staging System (ISS) consists of following 3 stages - Stage I: serum beta2-microglobulin less than (<) 3.5 milligrams per liter (mg/L) and albumin greater than or equal to (>=) 3.5 grams per 100 Milliliter (g/100 mL); Stage II: neither stage I nor stage III and Stage III: serum beta2-microglobulin >= 5.5 mg/L.
  Participants
    Stage I | 103 | 98 | 201
    Stage II | 156 | 163 | 319
    Stage III | 110 | 107 | 217
Time from Multiple Myeloma (MM) diagnosis [Mean (Standard Deviation); unit: Months] — Time from MM diagnosis is the time from diagnosis of multiple myeloma to randomization in each treatment group.
  Months | 1.3 (1.4) | 1.4 (1.5) | 1.3 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as time from date of randomization to either progressive disease (PD) or death, whichever occurred first based on computerized algorithm as per IMWG criteria. PD was defined as an increase of 25 percent (%) from the lowest response value in one of the following: serum and urine M-component (absolute increase must be greater than or equal to [>=] 0.5 gram per deciliter [g/dL] and >=200 milligram [mg]/24 hours respectively); Only in participants without measurable serum and urine M-protein levels the difference between involved and uninvolved free light chain (FLC) levels (absolute increase must be greater than [>]10 mg/dL); Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that could be attributed solely to Plasma cell (PC) proliferative disorder.
Time Frame: From randomization (Day -3) to disease progression, death, subsequent anti-myeloma therapy, withdrawal of consent to study participation or clinical cut-off (CCO) whichever occurs first (up to 3.5 years)
Population: Intent-to-treat (ITT) population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 369 | 368
Months | 31.87 [28.94 to NA] — Here NA signifies upper limit of confidence interval (CI) was not estimable due to an insufficient number of events. | NA [NA to NA] — Here 'NA' signifies median and CI was not estimable due to an insufficient number of events.
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.43 to 0.73]

2. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Better
Description: Percentage of participants with a CR or better (CR or stringent complete response [sCR]) based on computerized algorithm as per IMWG criteria was reported. CR was defined as negative immunofixation on the serum and urine, and disappearance of any soft tissue plasmacytomas, and less than (<) 5 percent (%) PCs in bone marrow. In participants with only measurable disease by serum FLC levels a normal serum FLC ratio was required. sCR was defined as in addition to CR a normal FLC ratio, and absence of clonal PCs by immunohistochemistry (IHC), immunofluorescence, 2-4 color flow cytometry (FC).
Time Frame: From randomization (Day -3) up to 6.6 years
Population: ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 369 | 368
Percentage of participants | 30.1 [25.4 to 35.0] | 51.1 [45.9 to 56.3]
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.44, 95% CI 2-sided [1.80 to 3.30]

3. Secondary Outcome: Percentage of Participants With Very Good Partial Response (VGPR) or Better
Description: VGPR or better rate was defined as the percentage of participants who achieved VGPR or better (VGPR, CR or sCR) according to the IMWG criteria during or after the study treatment. VGPR: Serum and urine component detectable by immunofixation but not on electrophoresis, or >= 90% reduction in serum M-protein plus urine M-protein level less than (<) 100 milligram (mg) per 24 hour; CR: negative immunofixation on the serum and urine, Disappearance of any soft tissue plasmacytomas and < 5% plasms cells (PCs) in bone marrow; sCR: CR in addition to having a normal FLC ratio and an absence of clonal cells in bone marrow by IHC, immunofluorescence, 2-4 color FC.
Time Frame: From randomization (Day -3) up to 6.6 years
Population: ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 369 | 368
Percentage of participants | 56.9 [51.7 to 62.0] | 81.5 [77.2 to 85.4]
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.4, 95% CI 2-sided [2.42 to 4.77]

4. Secondary Outcome: Percentage of Participants With Negative Minimal Residual Disease (MRD)
Description: MRD negativity rate is defined as the percentage of participants who had negative MRD at any time point after the date of randomization and prior to subsequent antimyeloma therapy. MRD was assessed in participants who achieved CR or better.
Time Frame: From randomization (Day -3) up to 6.6 years
Population: ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 369 | 368
Percentage of participants | 11.1 [8.1 to 14.8] | 32.1 [27.3 to 37.1]
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Test type: Superiority; p < 0.0001, Fisher Exact; Odds Ratio (OR) = 3.78, 95% CI 2-sided [2.55 to 5.59]

5. Secondary Outcome: Percentage of Participants With Stringent Complete Response (sCR)
Description: sCR as per IMWG criteria is CR plus normal free light chain (FLC) ratio and absence of clonal PCs by IHC, immunofluorescence or 2- to 4-color FC. CR: Negative immunofixation on the serum and urine; Disappearance of any soft tissue plasmacytomas; <5% PCs in bone marrow.
Time Frame: From randomization (Day -3) up to 6.6 years
Population: Intent-to-treat (ITT) population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 369 | 368
Percentage of participants | 15.7 [12.2 to 19.8] | 35.6 [30.7 to 40.7]
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.98, 95% CI 2-sided [2.09 to 4.24]

6. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was the percentage of participants who achieved partial response (PR) or better (PR, VGPR, CR or sCR) based on computerized algorithm as per IMWG criteria. PR: >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to <200 mg/24 hours. If serum and urine M-protein were not measurable, a decrease of >=50% in the difference between involved and uninvolved FLC levels was required in place of the M-protein criteria. If present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas was also required. VGPR: serum and urine M-component detectable by immunofixation but not on electrophoresis or >=90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours. CR: negative immunofixation on the serum and urine, Disappearance of any soft tissue plasmacytomas and < 5% PCs in bone marrow; sCR: CR in addition to having a normal FLC ratio and an absence of clonal cells in bone marrow by IHC, immunofluorescence, 2-4 color FC.
Time Frame: From randomization (Day -3) up to 6.6 years
Population: ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 369 | 368
Percentage of participants | 81.6 [77.2 to 85.4] | 92.9 [89.8 to 95.3]
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3, 95% CI 2-sided [1.85 to 4.86]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was measured from the date of randomization to the date of the death. Median OS was estimated by using the Kaplan-Meier method.
Time Frame: From randomization (Day -3) up to 8.7 years
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 369 | 368
Months | 64.07 [55.98 to 70.80] | 90.25 [80.76 to NA] — Here, 'NA' signifies that upper limit of 95% CI was not estimable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.55 to 0.82]

8. Secondary Outcome: Time to Disease Progression (TTP)
Description: TTP was defined as the time from the date of randomization to date of first documented evidence of PD or death due to PD, whichever occurred first. PD per IMWG criteria- Increase of 25 % from lowest response value in one of following: Serum M-component (absolute increase >=0.5 g/dL); Urine M-component (absolute increase >=200 mg/24 hours); Only in participants without measurable serum and urine M-protein levels: difference between involved and uninvolved FLC levels (absolute increase >10 milligram per deciliter [mg/dL]); Definite development of new bone lesions/soft tissue plasmacytomas or definite increase in size of existing bone lesions/soft tissue plasmacytomas and Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to the PC proliferative disorder.
Time Frame: From randomization (Day -3) up to 6.6 years
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 369 | 368
Months | 40.87 [35.81 to 48.79] | NA [NA to NA] — Here 'NA' signifies median, upper and lower limit of 95% CI was not estimable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.39 to 0.62]

9. Secondary Outcome: Time to Response
Description: Time to first response, time to VGPR or better, time to CR or better and time to best response was reported for this endpoint. Time to response: time from date of randomization to first efficacy evaluation that met criteria for PR/better as their best response (PR, CR, or better) based on IMWG criteria. PR: >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to <200 mg/24 hours. If serum and urine M-protein were not measurable, a decrease of >=50% in difference between involved and uninvolved FLC levels was required in place of M-protein criteria. Based on computerized algorithm, according to IMWG response criteria, VGPR or better: proportion of participants with a response of VGPR or better (i.e., VGPR, CR or sCR), CR or better: proportion of participants with a response of CR or better (i.e., CR or sCR).
Time Frame: From randomization (Day -3) up to 6.6 years
Population: Response evaluable population included all participants with confirmed diagnosis of multiple myeloma and measurable disease at baseline or screening visit and received at least one administration of study treatment and had adequate postbaseline disease assessments. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here 'n' signifies number of participants analyzed at specified timepoints.
Measure: Median (Full Range); unit: Months
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 301 | 342
Months
  Time to first response | 1.05 [0.3 to 22.3] | 1.05 [0.2 to 12.1]
  Time to VGPR or better: number analyzed (Participants) | 210 | 300
  Time to VGPR or better | 4.70 [0.9 to 43.3] | 3.01 [0.9 to 60.9]
  Time to CR or better: number analyzed (Participants) | 111 | 188
  Time to CR or better | 13.17 [2.8 to 54.6] | 10.66 [1.0 to 46.7]
  Time to best response | 6.31 [0.9 to 55.2] | 9.97 [0.9 to 60.9]

10. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined for participants with confirmed response (PR or better) as time between first documentation of response and disease progression per IMWG response criteria, or death due to PD, whichever occurs first. PD per IMWG criteria- Increase of 25 % from lowest response value in one of following: Serum M-component (absolute increase >=0.5 g/dL); Urine M-component (absolute increase >=200 mg/24 hours); Only in participants without measurable serum and urine M-protein levels: difference between involved and uninvolved FLC levels (absolute increase >10 milligram per deciliter [mg/dL]); Definite development of new bone lesions/soft tissue plasmacytomas or definite increase in size of existing bone lesions/soft tissue plasmacytomas and Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to the PC proliferative disorder.
Time Frame: From randomization (Day -3) up to 6.6 years
Population: Response evaluable population included all participants with confirmed diagnosis of multiple myeloma and measurable disease at baseline or screening visit and received at least one administration of study treatment and had adequate postbaseline disease assessments. Here, 'N' (Overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 152 | 119
Months | 43.7 [36.8 to 52.6] | NA [NA to NA] — Here 'NA' signifies median, upper and lower of 95% CI was not estimable due to an insufficient number of participants with events.

11. Secondary Outcome: Time to Subsequent Anti-myeloma Treatment
Description: Time to subsequent anti-myeloma treatment was defined as the time from randomization to the start of subsequent anti-myeloma treatment. Kaplan-Meier method was used for the analysis.
Time Frame: From randomization (Day -3) up to 8.7 years
Population: Intent-to-treat (ITT) population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 369 | 368
Months | 42.4 [33.5 to 50.6] | NA [84.1 to NA] — Here 'NA' signifies median and upper limit of 95% CI was not estimable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.41 to 0.63]

12. Secondary Outcome: Progression-free Survival on Next Line of Therapy (PFS2)
Description: PFS2 was defined as the time from randomization to progression on next line of therapy or death, whichever comes first. Disease progression on next line of treatment was based on investigator judgment.
Time Frame: From randomization (Day -3) up to 6.6 years
Population: Intent-to-treat (ITT) population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 369 | 368
Months | 48.89 [44.09 to 56.57] | 73.72 [73.72 to NA] — Here 'NA' signifies upper limit of 95% CI was not estimable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.49 to 0.76]

13. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C30 Global Health Status Score
Description: EORTC QLQ-C30 was 30 items self-reporting questionnaire, with 1 week recall period, resulting in 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 Global Health Status (GHS) scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Questionnaire included 28 items with 4-point Likert type responses from "1-not at all" to "4-very much" to assess functioning and symptoms; 2 items with 7-point Likert scales (1= poor and 7= excellent) for global health and overall health related QoL. Scores were transformed to 0 to 100 scale, with higher scores represented better GHS and functioning, and more symptoms. Negative change from baseline values showed deterioration in quality of life or functioning and reduction in symptom and positive values indicated improvement and worsening of symptoms.
Time Frame: Baseline (Day -24) and Day 1 of Cycles 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 and 66 (each Cycle of 28 days)
Population: ITT population included all randomized participants. Here 'N' (overall number of participants analyzed) signifies number of participants who were evaluable for this outcome measure; 'n' (number analyzed) signifies number of participants analyzed at specified timepoints.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 295 | 314
Score on scale
  Cycle 3 Day 1 | 1.4 [-0.7 to 3.5] | 3.8 [1.7 to 5.8]
  Cycle 6 Day 1: number analyzed (Participants) | 267 | 304
  Cycle 6 Day 1 | 4.8 [2.6 to 7] | 6.3 [4.3 to 8.4]
  Cycle 9 Day 1: number analyzed (Participants) | 229 | 278
  Cycle 9 Day 1 | 5.7 [3.4 to 8] | 7.5 [5.4 to 9.7]
  Cycle 12 Day 1: number analyzed (Participants) | 231 | 274
  Cycle 12 Day 1 | 4.5 [2.2 to 6.8] | 7.8 [5.6 to 9.9]
  Cycle 18 Day 1: number analyzed (Participants) | 186 | 253
  Cycle 18 Day 1 | 4.7 [2.2 to 7.2] | 6.4 [4.1 to 8.6]
  Cycle 24 Day 1: number analyzed (Participants) | 161 | 238
  Cycle 24 Day 1 | 4.7 [2.1 to 7.4] | 6.3 [4.1 to 8.6]
  Cycle 30 Day 1: number analyzed (Participants) | 140 | 213
  Cycle 30 Day 1 | 4.5 [1.7 to 7.3] | 5.5 [3.1 to 7.9]
  Cycle 36 Day 1: number analyzed (Participants) | 119 | 207
  Cycle 36 Day 1 | 5 [2 to 8] | 7.7 [5.3 to 10.1]
  Cycle 42 Day 1: number analyzed (Participants) | 100 | 184
  Cycle 42 Day 1 | 3.8 [0.6 to 7] | 5.6 [3.1 to 8.1]
  Cycle 48 Day 1: number analyzed (Participants) | 80 | 170
  Cycle 48 Day 1 | 3.4 [-0.1 to 6.9] | 4.2 [1.6 to 6.7]
  Cycle 54 Day 1: number analyzed (Participants) | 64 | 145
  Cycle 54 Day 1 | 6.1 [2.2 to 9.9] | 4.8 [2 to 7.5]
  Cycle 60 Day 1: number analyzed (Participants) | 46 | 114
  Cycle 60 Day 1 | 4.9 [0.4 to 9.4] | 4.1 [1.1 to 7.1]
  Cycle 66 Day 1: number analyzed (Participants) | 26 | 78
  Cycle 66 Day 1 | 7.1 [1.3 to 12.8] | 7.7 [4.2 to 11.2]
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); For Cycle 3 Day 1; Test type: Superiority; p = 0.0986, Mixed Models Analysis; Least Square Mean Difference = 2.4, 95% CI 2-sided [-0.4 to 5.2]
Statistical Analysis 2: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 6 Day 1; Test type: Superiority; p = 0.3042, Mixed Models Analysis; Least Square Mean Difference = 1.5, 95% CI 2-sided [-1.4 to 4.4]
Statistical Analysis 3: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 9 Day 1; Test type: Superiority; p = 0.2339, Mixed Models Analysis; Least Square Mean Difference = 1.8, 95% CI 2-sided [-1.2 to 4.9]
Statistical Analysis 4: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 12 Day 1; Test type: Superiority; p = 0.0365, Mixed Models Analysis; Least Square Mean Difference = 3.3, 95% CI 2-sided [0.2 to 6.3]
Statistical Analysis 5: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 18 Day 1; Test type: Superiority; p = 0.3093, Mixed Models Analysis — Cycle 24 Day 1; Least Square Mean Difference = 1.7, 95% CI 2-sided [-1.6 to 4.9]
Statistical Analysis 6: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 24 Day 1; Test type: Superiority; p = 0.3481, Mixed Models Analysis; Least Square Mean Difference = 1.6, 95% CI 2-sided [-1.8 to 5]
Statistical Analysis 7: Comparison: Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 30 Day 1; Test type: Superiority; p = 0.5825, Mixed Models Analysis; Least Square Mean Difference = 1, 95% CI 2-sided [-2.6 to 4.6]
Statistical Analysis 8: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 36 Day 1; Test type: Superiority; p = 0.1566, Mixed Models Analysis; Least Square Mean Difference = 2.7, 95% CI 2-sided [-1 to 6.4]
Statistical Analysis 9: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 42 Day 1; Test type: Superiority; p = 0.3858, Mixed Models Analysis; Least Square Mean Difference = 1.8, 95% CI 2-sided [-2.2 to 5.7]
Statistical Analysis 10: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 48 Day 1; Test type: Superiority; p = 0.7296, Least Square Mean Difference; Least Square Mean = 0.8, 95% CI 2-sided [-3.5 to 5]
Statistical Analysis 11: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 54 Day 1; Test type: Superiority; p = 0.5793, Mixed Models Analysis; Least Square Mean Difference = -1.3, 95% CI 2-sided [-6 to 3.3]
Statistical Analysis 12: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 60 Day 1; Test type: Superiority; p = 0.7756, Mixed Models Analysis; Least Square Mean Difference = -0.8, 95% CI 2-sided [-6.1 to 4.5]
Statistical Analysis 13: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 66 Day 1; Test type: Superiority; p = 0.8458, Mixed Models Analysis; Least Square Mean Difference = 0.7, 95% CI 2-sided [-6 to 7.4]

14. Secondary Outcome: Change From Baseline in EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) Visual Analogue Scale (VAS)
Description: EQ-5D-5L was a standardized, participant-rated questionnaire to assess health-related quality of life. The EQ-5D-5L includes 2 components: the EQ-5D-5L health state profile (descriptive system) and the EQ-5D-5L Visual Analog Scale. The Visual Analogue Scale was designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Time Frame: Baseline (Day -24) and Day 1 of Cycles 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 and 66 (each Cycle of 28 days)
Population: ITT population included all randomized participants. Here 'N' (overall number of participants analyzed) signifies number of participants who were evaluable for this outcome measure; 'n' signifies number of participants analyzed at specified timepoints.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 286 | 301
Score on scale
  Cycle 3 Day 1 | 2.1 [0.3 to 4] | 4.2 [2.3 to 6]
  Cycle 6 Day 1: number analyzed (Participants) | 252 | 287
  Cycle 6 Day 1 | 4.8 [2.8 to 6.8] | 7.6 [5.8 to 9.5]
  Cycle 9 Day 1: number analyzed (Participants) | 221 | 267
  Cycle 9 Day 1 | 7 [5 to 9.1] | 9.6 [7.7 to 11.5]
  Cycle 12 Day 1: number analyzed (Participants) | 227 | 261
  Cycle 12 Day 1 | 3.6 [1.6 to 5.7] | 9.4 [7.4 to 11.3]
  Cycle 18 Day 1: number analyzed (Participants) | 180 | 242
  Cycle 18 Day 1 | 5.4 [3.2 to 7.6] | 7.4 [5.4 to 9.4]
  Cycle 24 Day 1: number analyzed (Participants) | 154 | 227
  Cycle 24 Day 1 | 4.3 [2 to 6.7] | 7 [5 to 9]
  Cycle 30 Day 1: number analyzed (Participants) | 133 | 198
  Cycle 30 Day 1 | 4.6 [2.1 to 7] | 6.9 [4.8 to 9.1]
  Cycle 36 Day 1: number analyzed (Participants) | 115 | 195
  Cycle 36 Day 1 | 4.9 [2.3 to 7.5] | 8.1 [6 to 10.2]
  Cycle 42 Day 1: number analyzed (Participants) | 99 | 178
  Cycle 42 Day 1 | 4.6 [1.8 to 7.3] | 5.6 [3.4 to 7.8]
  Cycle 48 Day 1: number analyzed (Participants) | 79 | 162
  Cycle 48 Day 1 | 5.5 [2.4 to 8.5] | 6.7 [4.5 to 9]
  Cycle 54 Day 1: number analyzed (Participants) | 64 | 141
  Cycle 54 Day 1 | 3.4 [0.1 to 6.7] | 5.8 [3.4 to 8.2]
  Cycle 60 Day 1: number analyzed (Participants) | 44 | 112
  Cycle 60 Day 1 | 5.8 [1.9 to 9.6] | 5.2 [2.6 to 7.8]
  Cycle 66 Day 1: number analyzed (Participants) | 26 | 74
  Cycle 66 Day 1 | 6.9 [2 to 11.8] | 5.6 [2.5 to 8.7]
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 3 Day 1; Test type: Superiority; p = 0.1176, Mixed Models Analysis; Least Square Mean Difference = 2, 95% CI 2-sided [-0.5 to 4.5]
Statistical Analysis 2: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 6 Day 1; Test type: Superiority; p = 0.0336, Mixed Models Analysis; Least Square Mean Difference = 2.8, 95% CI 2-sided [0.2 to 5.4]
Statistical Analysis 3: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 9 Day 1; Test type: Superiority; p = 0.0653, Mixed Models Analysis; Least Square Mean Difference = 2.6, 95% CI 2-sided [-0.2 to 5.3]
Statistical Analysis 4: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 12 Day 1; Test type: Superiority; p = 0.0000, Mixed Models Analysis; Least Square Mean Difference = 5.8, 95% CI 2-sided [3 to 8.5]
Statistical Analysis 5: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 18 Day 1; Test type: Superiority; p = 0.1805, Mixed Models Analysis; Least Square Mean Difference = 2, 95% CI 2-sided [-0.9 to 4.8]
Statistical Analysis 6: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 24 Day 1; Test type: Superiority; p = 0.0783, Mixed Models Analysis; Least Square Mean Difference = 2.7, 95% CI 2-sided [-0.3 to 5.7]
Statistical Analysis 7: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 30 Day 1; Test type: Superiority; p = 0.1422, Mixed Models Analysis; Least Square Mean Difference = 2.4, 95% CI 2-sided [-0.8 to 5.5]
Statistical Analysis 8: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 36 Day 1; Test type: Superiority; p = 0.0575, Least Square Mean Difference; Least Square Mean = 3.2, 95% CI 2-sided [-0.1 to 6.5]
Statistical Analysis 9: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 42 Day 1; Test type: Superiority; p = 0.5339, Mixed Models Analysis; Least Square Mean Difference = 1.1, 95% CI 2-sided [-2.4 to 4.5]
Statistical Analysis 10: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 48 Day 1; Test type: Superiority; p = 0.5015, Mixed Models Analysis; Least Square Mean Difference = 1.3, 95% CI 2-sided [-2.4 to 5]
Statistical Analysis 11: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 54 Day 1; Test type: Superiority; p = 0.2512, Mixed Models Analysis; Least Square Mean Difference = 2.3, 95% CI 2-sided [-1.7 to 6.3]
Statistical Analysis 12: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 60 Day 1; Test type: Superiority; p = 0.8246, Mixed Models Analysis; Least Square Mean Difference = -0.5, 95% CI 2-sided [-5.1 to 4.1]
Statistical Analysis 13: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 66 Day 1; Test type: Superiority; p = 0.6640, Mixed Models Analysis; Least Square Mean Difference = -1.3, 95% CI 2-sided [-7 to 4.5]

15. Secondary Outcome: Change From Baseline in EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) Utility Score
Description: EQ-5D-5L was standardized, participant-reported questionnaire to assess health-related quality of life. EQ-5D-5L included 2 components: EQ-5D-5L health state profile (descriptive system) and EQ-5D-5L VAS. EQ-5D-5L descriptive system provided a profile of participant's health state 5 dimensions (5D): mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension had 5 response options (no problems, slight problems, moderate problems, severe problems and extreme problems) that reflected increasing levels of difficulty. Participants indicated their health state by selecting the most appropriate level in each of the 5D. Responses to the 5D scores were combined and converted into single preference-weighted health utility index score 0 (0.0- worst health state) to 1 (1.0- better health state) representing the general health status of individual (but allows for values less than 0 by United kingdom scoring algorithm). Higher score indicated better health state.
Time Frame: Baseline (Day -24) and Day 1 of Cycles 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 and 66 (each Cycle of 28 days)
Population: as for outcome 14
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 286 | 302
Score on scale
  Cycle 3 Day 1 | 0.081 [0.058 to 0.103] | 0.097 [0.074 to 0.119]
  Cycle 6 Day 1: number analyzed (Participants) | 252 | 287
  Cycle 6 Day 1 | 0.111 [0.087 to 0.135] | 0.13 [0.107 to 0.152]
  Cycle 9 Day 1: number analyzed (Participants) | 221 | 267
  Cycle 9 Day 1 | 0.113 [0.088 to 0.138] | 0.124 [0.101 to 0.147]
  Cycle 12 Day 1: number analyzed (Participants) | 227 | 261
  Cycle 12 Day 1 | 0.103 [0.078 to 0.128] | 0.132 [0.108 to 0.155]
  Cycle 18 Day 1: number analyzed (Participants) | 180 | 242
  Cycle 18 Day 1 | 0.089 [0.062 to 0.116] | 0.116 [0.092 to 0.14]
  Cycle 24 Day 1: number analyzed (Participants) | 154 | 227
  Cycle 24 Day 1 | 0.088 [0.059 to 0.116] | 0.121 [0.096 to 0.145]
  Cycle 30 Day 1: number analyzed (Participants) | 133 | 198
  Cycle 30 Day 1 | 0.088 [0.058 to 0.118] | 0.102 [0.076 to 0.127]
  Cycle 36 Day 1: number analyzed (Participants) | 115 | 195
  Cycle 36 Day 1 | 0.099 [0.067 to 0.131] | 0.109 [0.083 to 0.135]
  Cycle 42 Day 1: number analyzed (Participants) | 99 | 178
  Cycle 42 Day 1 | 0.062 [0.028 to 0.096] | 0.113 [0.086 to 0.14]
  Cycle 48 Day 1: number analyzed (Participants) | 79 | 162
  Cycle 48 Day 1 | 0.075 [0.038 to 0.112] | 0.082 [0.055 to 0.11]
  Cycle 54 Day 1: number analyzed (Participants) | 64 | 141
  Cycle 54 Day 1 | 0.05 [0.01 to 0.091] | 0.087 [0.058 to 0.116]
  Cycle 60 Day 1: number analyzed (Participants) | 44 | 112
  Cycle 60 Day 1 | 0.068 [0.02 to 0.115] | 0.079 [0.047 to 0.111]
  Cycle 66 Day 1: number analyzed (Participants) | 26 | 74
  Cycle 66 Day 1 | 0.041 [-0.019 to 0.102] | 0.111 [0.073 to 0.148]
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 3 Day 1; Test type: Superiority; p = 0.3069, Mixed Models Analysis; Least Square Mean Difference = 0.016, 95% CI 2-sided [-0.015 to 0.046]
Statistical Analysis 2: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 6 Day 1; Test type: Superiority; p = 0.2472, Mixed Models Analysis; Least Square Mean Difference = 0.019, 95% CI 2-sided [-0.013 to 0.05]
Statistical Analysis 3: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 9 Day 1; Test type: Superiority; p = 0.4972, Mixed Models Analysis; Least Square Mean Difference = 0.011, 95% CI 2-sided [-0.021 to 0.044]
Statistical Analysis 4: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 12 Day 1; Test type: Superiority; p = 0.0841, Mixed Models Analysis; Least Square Mean Difference = 0.029, 95% CI 2-sided [-0.004 to 0.062]
Statistical Analysis 5: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 18 Day 1; Test type: Superiority; p = 0.1296, Mixed Models Analysis; Least Square Mean Difference = 0.027, 95% CI 2-sided [-0.008 to 0.062]
Statistical Analysis 6: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 24 Day 1; Test type: Superiority; p = 0.0762, Mixed Models Analysis; Least Square Mean Difference = 0.033, 95% CI 2-sided [-0.003 to 0.07]
Statistical Analysis 7: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 30 Day 1; Test type: Superiority; p = 0.4859, Mixed Models Analysis; Least Square Mean Difference = 0.014, 95% CI 2-sided [-0.025 to 0.052]
Statistical Analysis 8: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 36 Day 1; Test type: Superiority; p = 0.6031, Mixed Models Analysis; Least Square Mean Difference = 0.011, 95% CI 2-sided [-0.029 to 0.051]
Statistical Analysis 9: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 42 Day 1; Test type: Superiority; p = 0.0178, Mixed Models Analysis; Least Square Mean Difference = 0.051, 95% CI 2-sided [0.009 to 0.093]
Statistical Analysis 10: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 48 Day 1; Test type: Superiority; p = 0.7460, Mixed Models Analysis; Least Square Mean Difference = 0.007, 95% CI 2-sided [-0.038 to 0.053]
Statistical Analysis 11: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 54 Day 1; Test type: Superiority; p = 0.1394, Mixed Models Analysis; Least Square Mean Difference = 0.037, 95% CI 2-sided [-0.012 to 0.086]
Statistical Analysis 12: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 60 Day 1; Test type: Superiority; p = 0.6982, Mixed Models Analysis; Least Square Mean Difference = 0.011, 95% CI 2-sided [-0.045 to 0.068]
Statistical Analysis 13: Comparison: Lenalidomide + Dexamethasone (Rd) vs Daratumumab + Lenalidomide + Dexamethasone (DRd); Cycle 66 Day 1; Test type: Superiority; p = 0.0543, Mixed Models Analysis; Least Square Mean Difference = 0.069, 95% CI 2-sided [-0.001 to 0.14]

16. Secondary Outcome: Sub-group Analysis: Progression-free Survival (PFS)
Description: PFS for participants with cytogenic high risk was reported. PFS was time from date of randomization to either PD or death, whichever occurred first based on computerized algorithm as per IMWG criteria. PD: an increase of 25% from lowest response value in one of following: serum and urine M-component (absolute increase must be >=0.5 g/dL and >=200 mg/24h respectively); Only in participants without measurable serum and urine M-protein levels, difference between involved and uninvolved FLC levels (absolute >10 mg/dL); Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in size of existing bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that could be attributed solely to PC proliferative disorder. High risk was defined as positive for any of del17p, t(14;16) or t(4;14) by (corrected serum calcium >11.5 mg/dL) Fluorescence In Situ Hybridization (FISH)/Karyotype.
Time Frame: From randomization (Day -3) to disease progression, death, subsequent anti-myeloma therapy, withdrawal of consent to study participation or clinical cut-off (CCO) whichever occurs first (up to 6.6 years).
Population: Intent-to-treat (ITT) population included all randomized participants. Here, 'N' signifies number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 31 | 28
Months | 29.6 [15.6 to 34.5] | 45.3 [18.4 to 61.9]

17. Secondary Outcome: Sub-group Analysis: Overall Response Rate (ORR)
Description: ORR for participants with cytogenic high risk was reported. ORR: percentage of participants who achieved PR/better per IMWG criteria. PR: >=50% reduction of serum M-protein, reduction in 24h urinary M-protein by >=90% or <200mg/24h. If serum/urine M-protein were not measurable, decrease of >=50% in difference between involved and uninvolved FLC levels was required in place of M-protein criteria. If present at baseline, >=50% reduction in size of soft tissue plasmacytomas was required. VGPR: serum/urine M-component detectable by immunofixation but not on electrophoresis or >=90% reduction in serum and urine M-protein <100mg/24h. CR: negative immunofixation on serum/urine, disappearance of soft tissue plasmacytomas, <5% PCs in bone marrow; sCR: CR in addition to normal FLC ratio, absence of clonal cells in bone marrow by IHC, immunofluorescence, 2-4 color FC. High risk: positive for any of del17p, t(14;16) or t(4;14) by FISH/Karyotype.
Time Frame: From randomization (Day -3) up to 6.6 years
Population: as for outcome 16
Measure: Number; unit: Percentage of participants
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
Number analyzed (Participants) | 44 | 48
Percentage of participants | 75.0 | 91.7

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization (Day -3) up to 8.7 years; Serious and Other AEs: From start of treatment (Day 1) up to 6.6 years
Description: Serious and Other AEs: Safety population was defined as participants who have received at least 1 administration of any study treatment (partial or complete).
Arm/Group | Lenalidomide + Dexamethasone (Rd) | Daratumumab + Lenalidomide + Dexamethasone (DRd)
All-Cause Mortality (participants affected / at risk) | 259/369 | 287/368
Serious Adverse Events (participants affected / at risk) | 262/365 | 289/364
Other Adverse Events (participants affected / at risk) | 358/365 | 362/364
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide + Dexamethasone (Rd) (N=365) | Daratumumab + Lenalidomide + Dexamethasone (DRd) (N=364)
Anaemia (Blood and lymphatic system disorders) | 12 | 6
Anaemia Macrocytic (Blood and lymphatic system disorders) | 1 | 0
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 | 0
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 9 | 11
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Acute Coronary Syndrome (Cardiac disorders) | 5 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 3
Angina Pectoris (Cardiac disorders) | 0 | 2
Arrhythmia (Cardiac disorders) | 1 | 0
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 15 | 10
Atrial Flutter (Cardiac disorders) | 3 | 3
Atrial Tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular Block (Cardiac disorders) | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 3 | 0
Cardiac Amyloidosis (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 4 | 3
Cardiac Failure (Cardiac disorders) | 11 | 5
Cardiac Failure Acute (Cardiac disorders) | 0 | 1
Cardiac Failure Chronic (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 5 | 3
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Cardiogenic Shock (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 2 | 3
Coronary Artery Stenosis (Cardiac disorders) | 0 | 1
Hypertensive Heart Disease (Cardiac disorders) | 0 | 1
Mitral Valve Incompetence (Cardiac disorders) | 0 | 2
Myocardial Infarction (Cardiac disorders) | 5 | 2
Myocardial Ischaemia (Cardiac disorders) | 1 | 2
Myocarditis (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 2
Sinus Node Dysfunction (Cardiac disorders) | 0 | 2
Sinus Tachycardia (Cardiac disorders) | 0 | 1
Stress Cardiomyopathy (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 1 | 1
Corneal Dystrophy (Congenital, familial and genetic disorders) | 0 | 1
Deafness Bilateral (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 2
Adrenal Insufficiency (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Blepharitis (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 5 | 4
Retinal Artery Occlusion (Eye disorders) | 0 | 1
Retinal Detachment (Eye disorders) | 1 | 0
Retinal Vein Thrombosis (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 3
Anal Fissure (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 5 | 2
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 2 | 4
Dental Caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 11
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 1 | 0
Diverticular Perforation (Gastrointestinal disorders) | 2 | 5
Diverticulum (Gastrointestinal disorders) | 1 | 0
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enterovesical Fistula (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 2 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 4 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 2 | 8
Inguinal Hernia Strangulated (Gastrointestinal disorders) | 1 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 1 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 3
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 1
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 2
Melaena (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 5
Obstruction Gastric (Gastrointestinal disorders) | 0 | 1
Obstructive Pancreatitis (Gastrointestinal disorders) | 0 | 1
Oesophageal Achalasia (Gastrointestinal disorders) | 0 | 1
Oesophageal Rupture (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 3
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 3
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 2 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2
Subileus (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 6
Asthenia (General disorders) | 6 | 6
Chest Discomfort (General disorders) | 1 | 0
Chest Pain (General disorders) | 3 | 0
Chills (General disorders) | 0 | 1
Extravasation (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 4
General Physical Health Deterioration (General disorders) | 12 | 3
Granuloma (General disorders) | 0 | 1
Influenza Like Illness (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 2 | 2
Non-Cardiac Chest Pain (General disorders) | 5 | 7
Oedema Peripheral (General disorders) | 0 | 2
Pain (General disorders) | 1 | 0
Peripheral Swelling (General disorders) | 0 | 1
Physical Deconditioning (General disorders) | 2 | 0
Procedural Failure (General disorders) | 1 | 0
Pyrexia (General disorders) | 12 | 20
Sudden Cardiac Death (General disorders) | 1 | 0
Sudden Death (General disorders) | 3 | 1
Systemic Inflammatory Response Syndrome (General disorders) | 1 | 0
Acute Hepatic Failure (Hepatobiliary disorders) | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 3 | 3
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 6
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 1 | 0
Hepatocellular Injury (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Amyloidosis (Immune system disorders) | 0 | 1
Abdominal Sepsis (Infections and infestations) | 1 | 0
Anal Abscess (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 0 | 2
Appendicitis Perforated (Infections and infestations) | 1 | 0
Arthritis Bacterial (Infections and infestations) | 1 | 0
Arthritis Infective (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 3
Bacterial Diarrhoea (Infections and infestations) | 0 | 1
Bacterial Sepsis (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 6 | 15
Campylobacter Gastroenteritis (Infections and infestations) | 1 | 0
Campylobacter Infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 4 | 5
Clostridium Difficile Colitis (Infections and infestations) | 1 | 3
Colonic Abscess (Infections and infestations) | 0 | 1
Coronavirus Infection (Infections and infestations) | 0 | 1
Covid-19 (Infections and infestations) | 0 | 6
Covid-19 Pneumonia (Infections and infestations) | 0 | 3
Cystitis (Infections and infestations) | 0 | 1
Cytomegalovirus Infection (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 4 | 7
Encephalitis Viral (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Endocarditis Staphylococcal (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 4 | 5
Escherichia Bacteraemia (Infections and infestations) | 0 | 1
Escherichia Pyelonephritis (Infections and infestations) | 1 | 0
Escherichia Sepsis (Infections and infestations) | 2 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal Viral Infection (Infections and infestations) | 1 | 0
Groin Abscess (Infections and infestations) | 2 | 1
Haematoma Infection (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1
Infected Cyst (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 8 | 17
Kidney Infection (Infections and infestations) | 0 | 1
Klebsiella Bacteraemia (Infections and infestations) | 1 | 1
Klebsiella Sepsis (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Listeriosis (Infections and infestations) | 0 | 1
Localised Infection (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 12 | 11
Lower Respiratory Tract Infection Bacterial (Infections and infestations) | 2 | 0
Lower Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0
Metapneumovirus Infection (Infections and infestations) | 1 | 1
Myocarditis Infectious (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Neutropenic Infection (Infections and infestations) | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 1 | 2
Nocardiosis (Infections and infestations) | 0 | 1
Oesophageal Candidiasis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 2 | 1
Otitis Externa (Infections and infestations) | 1 | 0
Parainfluenzae Virus Infection (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pleural Infection (Infections and infestations) | 0 | 1
Pneumocystis Jirovecii Infection (Infections and infestations) | 0 | 1
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 39 | 68
Pneumonia Bacterial (Infections and infestations) | 1 | 1
Pneumonia Klebsiella (Infections and infestations) | 0 | 1
Pneumonia Pneumococcal (Infections and infestations) | 1 | 0
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 0 | 1
Pulmonary Mycosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 3
Pyelonephritis Acute (Infections and infestations) | 0 | 1
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 1 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 2 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 3
Salmonellosis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 10 | 11
Sepsis Syndrome (Infections and infestations) | 0 | 1
Septic Arthritis Staphylococcal (Infections and infestations) | 0 | 1
Septic Embolus (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 3 | 6
Skin Infection (Infections and infestations) | 0 | 1
Soft Tissue Infection (Infections and infestations) | 1 | 0
Spinal Cord Infection (Infections and infestations) | 1 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 1 | 1
Streptococcal Sepsis (Infections and infestations) | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 6
Ureteritis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 7 | 12
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 3
Varicella (Infections and infestations) | 0 | 1
Varicella Zoster Virus Infection (Infections and infestations) | 1 | 0
Vascular Device Infection (Infections and infestations) | 0 | 2
Vestibular Neuronitis (Infections and infestations) | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Vulval Abscess (Infections and infestations) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0
Acetabulum Fracture (Injury, poisoning and procedural complications) | 0 | 1
Animal Bite (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous Fistula Site Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 1
Face Injury (Injury, poisoning and procedural complications) | 0 | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 6 | 9
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 4 | 6
Femur Fracture (Injury, poisoning and procedural complications) | 5 | 9
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Head Injury (Injury, poisoning and procedural complications) | 1 | 3
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 5
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 2
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0
Limb Injury (Injury, poisoning and procedural complications) | 2 | 0
Limb Traumatic Amputation (Injury, poisoning and procedural complications) | 0 | 1
Open Fracture (Injury, poisoning and procedural complications) | 1 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 2 | 2
Periorbital Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Periprosthetic Fracture (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Fever (Injury, poisoning and procedural complications) | 1 | 0
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 3
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 4 | 6
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 1
Sternal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 3
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Ulna Fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 2
Wound Necrosis (Injury, poisoning and procedural complications) | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Blood Creatinine Increased (Investigations) | 2 | 0
C-Reactive Protein Increased (Investigations) | 1 | 2
General Physical Condition Abnormal (Investigations) | 0 | 1
International Normalised Ratio Increased (Investigations) | 1 | 0
Lipase Increased (Investigations) | 0 | 1
Occult Blood Positive (Investigations) | 1 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 1
Radial Pulse Abnormal (Investigations) | 1 | 0
Transaminases Increased (Investigations) | 2 | 0
Troponin I Increased (Investigations) | 1 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 6
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 1
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 | 1
Failure to Thrive (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 3 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 14
Bone Lesion (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Bone Sequestrum (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 1
Crystal Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral Disc Compression (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Jaw Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 5
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 4
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 2 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B Precursor Type Acute Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Gastrointestinal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive Lobular Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mantle Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mucinous Adenocarcinoma of Appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine Carcinoma of the Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Porocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Primary Pulmonary Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin Squamous Cell Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 7
Superficial Spreading Melanoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Balance Disorder (Nervous system disorders) | 1 | 1
Brain Oedema (Nervous system disorders) | 1 | 0
Brain Stem Infarction (Nervous system disorders) | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 3 | 1
Cerebral Ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 5 | 5
Cognitive Disorder (Nervous system disorders) | 0 | 3
Dementia (Nervous system disorders) | 0 | 1
Dementia Alzheimer's Type (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 3
Encephalopathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Focal Dyscognitive Seizures (Nervous system disorders) | 0 | 1
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 1
Haemorrhagic Stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hepatic Encephalopathy (Nervous system disorders) | 0 | 2
Hyperaesthesia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Ischaemic Cerebral Infarction (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 3 | 2
Nervous System Disorder (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 1
Occipital Neuralgia (Nervous system disorders) | 1 | 0
Orthostatic Intolerance (Nervous system disorders) | 0 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1
Post Herpetic Neuralgia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 2 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 2 | 4
Seizure (Nervous system disorders) | 2 | 5
Spinal Cord Compression (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 4 | 6
Transient Ischaemic Attack (Nervous system disorders) | 3 | 2
Vertebrobasilar Stroke (Nervous system disorders) | 1 | 0
Vith Nerve Paralysis (Nervous system disorders) | 1 | 0
Device Dislocation (Product Issues) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Completed Suicide (Psychiatric disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 3 | 4
Depression (Psychiatric disorders) | 1 | 1
Eating Disorder (Psychiatric disorders) | 1 | 0
Major Depression (Psychiatric disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 2 | 3
Personality Change (Psychiatric disorders) | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 15 | 14
Bladder Neck Sclerosis (Renal and urinary disorders) | 0 | 1
Bladder Stenosis (Renal and urinary disorders) | 0 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 2
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 1
Renal Disorder (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 5 | 6
Renal Impairment (Renal and urinary disorders) | 2 | 0
Urethral Caruncle (Renal and urinary disorders) | 0 | 1
Urethral Stenosis (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 5 | 2
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 3
Cystocele (Reproductive system and breast disorders) | 1 | 0
Genital Prolapse (Reproductive system and breast disorders) | 1 | 1
Hysterocele (Reproductive system and breast disorders) | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Bronchial Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 14 | 16
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute Febrile Neutrophilic Dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis Exfoliative Generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Drug Reaction with Eosinophilia and Systemic Symptoms (Skin and subcutaneous tissue disorders) | 4 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Air Embolism (Vascular disorders) | 0 | 1
Aortic Aneurysm (Vascular disorders) | 0 | 1
Aortic Aneurysm Rupture (Vascular disorders) | 1 | 0
Aortic Stenosis (Vascular disorders) | 1 | 0
Arteritis (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 10 | 6
Embolism (Vascular disorders) | 1 | 2
Haematoma (Vascular disorders) | 4 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 1 | 3
Orthostatic Hypotension (Vascular disorders) | 1 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 0
Peripheral Artery Stenosis (Vascular disorders) | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 0 | 2
Phlebitis (Vascular disorders) | 2 | 1
Superior Vena Cava Occlusion (Vascular disorders) | 0 | 1
Venous Thrombosis (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide + Dexamethasone (Rd) (N=365) | Daratumumab + Lenalidomide + Dexamethasone (DRd) (N=364)
Anaemia (Blood and lymphatic system disorders) | 148 | 154
Leukopenia (Blood and lymphatic system disorders) | 42 | 73
Lymphopenia (Blood and lymphatic system disorders) | 48 | 72
Neutropenia (Blood and lymphatic system disorders) | 167 | 224
Thrombocytopenia (Blood and lymphatic system disorders) | 76 | 82
Atrial Fibrillation (Cardiac disorders) | 33 | 30
Vertigo (Ear and labyrinth disorders) | 19 | 22
Cataract (Eye disorders) | 78 | 88
Vision Blurred (Eye disorders) | 19 | 30
Abdominal Pain (Gastrointestinal disorders) | 43 | 59
Abdominal Pain Upper (Gastrointestinal disorders) | 30 | 41
Constipation (Gastrointestinal disorders) | 136 | 156
Diarrhoea (Gastrointestinal disorders) | 186 | 237
Dry Mouth (Gastrointestinal disorders) | 21 | 14
Dyspepsia (Gastrointestinal disorders) | 31 | 31
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 24 | 24
Haemorrhoids (Gastrointestinal disorders) | 11 | 19
Nausea (Gastrointestinal disorders) | 87 | 133
Stomatitis (Gastrointestinal disorders) | 13 | 25
Toothache (Gastrointestinal disorders) | 20 | 20
Vomiting (Gastrointestinal disorders) | 48 | 77
Asthenia (General disorders) | 99 | 134
Chills (General disorders) | 6 | 49
Fatigue (General disorders) | 114 | 163
Influenza Like Illness (General disorders) | 17 | 22
Non-Cardiac Chest Pain (General disorders) | 21 | 23
Oedema Peripheral (General disorders) | 117 | 156
Peripheral Swelling (General disorders) | 24 | 16
Pyrexia (General disorders) | 63 | 85
Hypogammaglobulinaemia (Immune system disorders) | 3 | 19
Bronchitis (Infections and infestations) | 85 | 119
Cystitis (Infections and infestations) | 10 | 23
Gastroenteritis (Infections and infestations) | 22 | 36
Influenza (Infections and infestations) | 22 | 31
Lower Respiratory Tract Infection (Infections and infestations) | 18 | 21
Nasopharyngitis (Infections and infestations) | 66 | 92
Pneumonia (Infections and infestations) | 36 | 64
Rhinitis (Infections and infestations) | 23 | 38
Sinusitis (Infections and infestations) | 17 | 26
Upper Respiratory Tract Infection (Infections and infestations) | 52 | 93
Urinary Tract Infection (Infections and infestations) | 44 | 77
Contusion (Injury, poisoning and procedural complications) | 32 | 37
Fall (Injury, poisoning and procedural complications) | 25 | 43
Alanine Aminotransferase Increased (Investigations) | 15 | 21
Blood Alkaline Phosphatase Increased (Investigations) | 9 | 20
Blood Creatinine Increased (Investigations) | 21 | 35
Weight Decreased (Investigations) | 70 | 115
Weight Increased (Investigations) | 8 | 29
Decreased Appetite (Metabolism and nutrition disorders) | 65 | 93
Dehydration (Metabolism and nutrition disorders) | 18 | 23
Gout (Metabolism and nutrition disorders) | 17 | 19
Hyperglycaemia (Metabolism and nutrition disorders) | 28 | 54
Hyperkalaemia (Metabolism and nutrition disorders) | 10 | 19
Hypocalcaemia (Metabolism and nutrition disorders) | 35 | 59
Hypokalaemia (Metabolism and nutrition disorders) | 72 | 100
Hypomagnesaemia (Metabolism and nutrition disorders) | 32 | 30
Hyponatraemia (Metabolism and nutrition disorders) | 16 | 20
Hypophosphataemia (Metabolism and nutrition disorders) | 10 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 78 | 107
Back Pain (Musculoskeletal and connective tissue disorders) | 107 | 147
Bone Pain (Musculoskeletal and connective tissue disorders) | 35 | 42
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 86 | 111
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 25 | 40
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 45 | 39
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 57 | 73
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 34
Neck Pain (Musculoskeletal and connective tissue disorders) | 33 | 31
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 21 | 30
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 60 | 82
Spinal Pain (Musculoskeletal and connective tissue disorders) | 19 | 17
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 22
Dizziness (Nervous system disorders) | 65 | 79
Dysgeusia (Nervous system disorders) | 17 | 29
Headache (Nervous system disorders) | 43 | 79
Hypoaesthesia (Nervous system disorders) | 17 | 23
Memory Impairment (Nervous system disorders) | 11 | 20
Paraesthesia (Nervous system disorders) | 31 | 67
Peripheral Sensory Neuropathy (Nervous system disorders) | 66 | 111
Sciatica (Nervous system disorders) | 19 | 26
Taste Disorder (Nervous system disorders) | 19 | 14
Tremor (Nervous system disorders) | 53 | 64
Agitation (Psychiatric disorders) | 10 | 20
Anxiety (Psychiatric disorders) | 38 | 39
Confusional State (Psychiatric disorders) | 20 | 29
Depression (Psychiatric disorders) | 38 | 37
Insomnia (Psychiatric disorders) | 116 | 125
Acute Kidney Injury (Renal and urinary disorders) | 17 | 34
Chronic Kidney Disease (Renal and urinary disorders) | 23 | 37
Dysuria (Renal and urinary disorders) | 11 | 20
Haematuria (Renal and urinary disorders) | 5 | 19
Renal Impairment (Renal and urinary disorders) | 35 | 34
Cough (Respiratory, thoracic and mediastinal disorders) | 65 | 123
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 19 | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 64 | 115
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 25 | 29
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 | 21
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 23
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 10 | 31
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 23
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12 | 30
Dry Skin (Skin and subcutaneous tissue disorders) | 21 | 30
Erythema (Skin and subcutaneous tissue disorders) | 22 | 31
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 23
Night Sweats (Skin and subcutaneous tissue disorders) | 20 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 35 | 41
Rash (Skin and subcutaneous tissue disorders) | 70 | 72
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 10 | 23
Skin Lesion (Skin and subcutaneous tissue disorders) | 9 | 19
Deep Vein Thrombosis (Vascular disorders) | 30 | 32
Haematoma (Vascular disorders) | 23 | 31
Hypertension (Vascular disorders) | 31 | 65
Hypotension (Vascular disorders) | 33 | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT02252172/Prot_002.pdf
  • Statistical Analysis Plan (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT02252172/SAP_003.pdf